CLINICAL TRIAL: NCT01578213
Title: Validation of Digital-PCR Analysis Through Programmed Imatinib Interruption in PCR Negative CML Patients (ISAV)
Brief Title: Validation of Digital-PCR Analysis Through Programmed Imatinib Interruption in PCR Negative CML Patients
Acronym: ISAV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ISAV; 2011-002749-37 (EudraCT Number)
Record Dates: First submitted 2012-04-13; First posted 2012-04-16 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib (Experimental)
  Interventions: Drug: Imatinib mesylate

INTERVENTIONS:
Drug: Imatinib mesylate — * Capsules, hard 50 or 100 mg/Film-coated Tablets 100 or 400 mg
  * Total dosage per day: 800 mg
  * Oral use
  Other Names: Glivec, Gleevec

SUMMARY:
The purpose of this study is to assess the capability of the dPCR technique to predict the absence of disease relapses after imatinib discontinuation in CML patients with negative Q-RT-PCR results for longer than 18 months.

DETAILED DESCRIPTION:
This study will recruit approximately 100 CML patients under imatinib therapy in complete molecular remission with a history of at least 18 months of consecutive negative standard Q-RT-PCR as performed in their own centers. After signing the informed consent form (ICF), the patients will be tested for dPCR and will discontinue imatinib therapy. Then they will be monitored by standard Q-RT-PCR to assess the maintenance of the molecular remission; collection of data will be prospective as each center will collect the data for 36 months. At the end of this period, a peripheral blood sample for dPCR analysis will be obtained from those patients who will still have undetectable BCR-ABL transcripts by Q-RT-PCR to verify CML eradication. The maintenance of molecular remission by Q-RT-PCR and the survival will be monitored every six months during an additional follow-up of 24 months. Patients found to be positive to BCR-ABL transcripts by standard Q-RTPCR will repeat the test every 2 to 4 weeks until the loss of molecular remission, defined as two consecutive BCR-ABL positive tests with at least one with BCR-ABL/BCR value above 0.1%, or until the end of the study, whichever come first.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated IRB/IEC-approved Informed Consent
2. Age>=18 years
3. Male or female patients with CML diagnosed in chronic or accelerated phase and who have been treated for more than 2 consecutive years with imatinib therapy
4. Sustained Complete Molecular Response (as defined by the treating center) for at least 18 months with imatinib treatment
5. A minimum of 3 CMR determined by Q-RT-PCR analysis to support disease status, with the list one performed within 3 calendar months prior to enrollment date
6. Willingness and ability to comply with scheduled visits laboratory tests and other study procedures

Exclusion Criteria:

1. Allogenic hematopoietic stem cell transplantation
2. Known active infections including human immunodeficiency virus (HIV) positivity
3. Current enrollment another clinical trial
4. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2011-11-09; Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
The Negative Predicted Value Ratio (rNPV) of dPCR over Q-RT-PCR | At 36 months.
  The capability of the dPCR method to predict relapse-free patients relative to the standard method. NPV of each method will be computed as the number of patients who are negative according to either method at the time of imatinib discontinuation and remain relapse-free 36 months later over the total of negative patients according to either method, respectively

SECONDARY OUTCOMES:
Rate of molecular and cytogenetic relapse | At 36 months
  Rate of molecular and cytogenetic relapse after discontinuation of imatinib treatment out of total number of patients enrolled
Rate of dPCR positive patients | At 36 months
  Rate of patients who are dPCR positive before discontinuation of imatinib and who do not relapse within the following 36 months (false positive) out of the total number of relapse-free patients at month 36.
Rate of dPCR negative patients | At 36 months
  Rate of patients who are dPCR negative before discontinuation of imatinib and who relapse (false negative) out of the total number of patients relapsing within the following 36 months.
Rate of patients who are maintaining dPCR negativity for 36 months | At 36 months
  Rate of patients who are maintaining dPCR negativity for 36 months over the patients who are Q-RT-PCR negative at the end of the interval.
Time to molecular relapse | At 36 months
  Time to molecular relapse, both from the first PCR-negative and from the discontinuation of imatinib to the time of loss of molecular response, respectively.
Overall Survival | At the end of the study
  Overall Survival
Quality of Life Assessment | At 36 months
  Quality of Life, as measured by the Global Health Status\QOL and other subscales scores of EORTC-QLQ-C30 questionnaire
Rate of patients progressing or developing resistance | At 36 months
  Rate of patients progressing or developing resistance after imatinib resumption out of total number of patients enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gambacorti-Passerini, MD, Study Director — Azienda Ospedaliera San Gerardo di Monza; Eros Di Bona, MD, Principal Investigator — Ospedale S. Bortolo (USSL 6); Francesco Di Raimondo, MD, Principal Investigator — Azienda Ospedaliero-Universitaria "Policlinico - Vittorio Emanuele"; Elisabetta Abruzzese, MD, Principal Investigator — Università di Tor Vergata Ospedale di S. Eugenio; Luca Arcaini, MD, Principal Investigator — IRCCS Policlinico San Matteo Pavia; Valeria Santini, MD, Principal Investigator — Università di Firenze Azienda Ospedaliera-Universitaria Careggi; Bruno Martino, MD, Principal Investigator — A.O. Bianchi-Melacrino-Morelli; Alessandra Iurlo, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico; Arnon Nagler, MD, Principal Investigator — Chaim Sheba Medical Center; Ester Pungolino, MD, Principal Investigator — Ospedale Niguarda Ca' Granda; Philipp le Coutre, MD, Principal Investigator — Charité University of Berlin; Sarit Assouline, MD, Principal Investigator — McGill University - Jewish General Hospital; Onno Leeskma, MD, Principal Investigator — Onze Lieve Vrouwe Gasthuis; Marcio Andrade, MD, Principal Investigator — Hospital Miguel Servet; Micaela Bergamaschi, MD, Principal Investigator — IRCCS A.O.U. San Martino
Locations (14):
- McGill University - Jewish General Hospital Division of Hematology and Department of Oncology, Montreal, Quebec, Canada
- Charité University of Berlin - Clinic of Medicine - Hematology and Oncology, Berlin, Germany
- Chaim Sheba Medical Center - Division of Hematology, BMT and CBB, Tel Litwinsky, Israel
- Italy (10):
  - Azienda Ospedaliero-Universitaria "Policlinico-Vittorio Emanuele", Catania, Italy/Catania
  - Università di Firenze Azienda Ospedaliera - Universitaria Careggi, Florence, Italy/Firenze
  - Azienda Ospedaliera San Gerardo di Monza, Monza, Italy/MB
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC di Ematologia, Milan, Italy/Milano
  - IRCCS Policlinico San Matteo Pavia - Istituto di Ematologia, Pavia, Italy/Pavia
  - A.O. Bianchi-Melacrino-Morelli U.O. Ematologia, Reggio Calabria, Italy/Reggio Calabria
  - Universita di Tor Vergata Ospedale S. Eugenio, Rome, Italy/Rome
  - Ospedale S. Bortolo (USSL 6), Vicenza, Italy/Vicenza
  - Ospedale Niguarda Ca' Granda - U.O. Ematologia, Milan, MI
  - IRCCS A.O.U. San Martino, Genova
- Hospital Universitario Miguel Servet - Hematologia, Zaragoza, Spain